CLINICAL TRIAL: NCT02455947
Title: The Effect of Inquiry Based Stress Reduction (IBSR) Meditation Technique on Levels of Burnout and Wellbeing Among Teachers.
Brief Title: IBSR Meditation Technique for Teachers' Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv Medical Center (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Shahar Lev- Ari, PhD, Dr. Shahar Lev-Ari, PhD, LLb, Tel Aviv Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TelAvivMC
Record Dates: First submitted 2015-05-20; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Burnout, Professional
Keywords: Burnout; Teachers; Meditation; IBSR; "The Work"; Byron Katie
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inquiry Based Stress Reduction (IBSR) (Experimental): IBSR intervention is the clinical implementation of a mindful-process, named "The Work" developed by Byron Katie.It teaches the individual to identify and question the thoughts that causes stress and suffering through four questions and turnarounds.
  Interventions: Other: Inquiry Based Stress Reduction (IBSR)
- Control group (No Intervention): A non interventional group/ The participants completed questionnaires before and after the intervention.

INTERVENTIONS:
Other: Inquiry Based Stress Reduction (IBSR) — During a 12-week intervention program, participants will be encouraged to identify and inquire their stressful thoughts.All the sessions were standardized according to a training manual, and were assessed after each session for maintaining consistency in the program.
  Other Names: The Work
  Arms: Inquiry Based Stress Reduction (IBSR)

SUMMARY:
The purpose of this study is to investigate the effect of Inquiry based stress reduction (IBSR) meditation technique on levels of burnout and wellbeing among teachers.

DETAILED DESCRIPTION:
Teachers' burnout is a well-known phenomenon with personal and professional implications. The current study investigates the effect of inquiry based stress reduction (IBSR) technique on burnout and well-being among teachers.

ELIGIBILITY:
Inclusion Criteria:

* All the teachers working in 'Begin' high-school, Rosh Hayin, Israel
* agreed to sign an informed consent form

Exclusion Criteria:

* Teachers with previous experience with IBSR technique

Ages: 20 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Burnout levels, Maslach Burnout Inventory (MBI) | 3 months
  emotional exhaustion and personal accomplishment

SECONDARY OUTCOMES:
Positive and Negative Affect Scale (PANAS) | 3 months
  Positive and Negative emotions at daily life
Depression, Anxiety, Stress (DASS) | 3 months
  Clinical psycological symptoms
Perceived Stress Scale (PSS ) | 3 months
  Stress levels at daily life

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Lev-Ari, PhD, Principal Investigator — Integartive Medicine, Tel Aviv Medical Center